CLINICAL TRIAL: NCT02277080
Title: The Immune and Endocrine Systems in Chronic Non-cancer Patients Treated With Opioids: Effects on Cognition, Pain and Quality of Life
Brief Title: The Immune and Endocrine Systems in Chronic Non-cancer Patients Treated With Opioids
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Per Sjogren, Professor, M.D., Dr. Med. Sci, Rigshospitalet, Denmark
Other Study IDs: H-1-2014-063
Record Dates: First submitted 2014-10-22; First posted 2014-10-28 (Estimated); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Pain; Opioids; Immune System; Endocrine System; Quality of Life
Keywords: Pain, opioids, immune system, endocrine system, quality of life
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood/serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Opioid group: These patients should have been treated only with one opioid (morphine, oxycodone, fentanyl, methadone, hydromorphone, tapentadol or tramadol) for more than one month
- Control group: Chronic non-cancer pain patients not treated with analgesics

SUMMARY:
The primary aim is to investigate the dose and time dependent effects of different opioids on the immune and endocrine systems.

The secondary aim is to investigate whether associations between the function of the immune and endocrine systems and opioid use influence cognitive function, pain and quality of life.

DETAILED DESCRIPTION:
BACKGROUND

Epidemiological data from the US and Denmark have shown that 3-5% of the population use opioids for treatment of chronic pain conditions.

Long-term use of opioids may cause "classic" opioid-induced adverse effects, but also serious consequences such as hyperalgesia, cognitive disorders, and suppression of the immune and endocrine systems.

Relatively few studies suggest that these substances affect hormone function in humans. The best studied is the circumstances regarding sex hormones.

A single systematic study and several clinical observations suggest that both pituitary-adrenal function and formation of growth hormone is also reduced by opioids.

Other studies have shown that not only are hormones changing during treatment with opioids, but the immunological function is also affected. There have been shown a link between the immunological and hormonal function so that parts of the immune system also affect the pituitary-adrenal function.

Opioid use and misuse per se has long been suspected to be associated with infections because both the innate and the adaptive immune system are getting affected through a number of mechanisms.

This study investigates the possibility of hormonal disorders being contributing factor to the development of cognitive impairment in patients who are in opioid treatment. The same applies to patients' well-being, mood and pain perception.

STUDY DESIGN

A cross-sectional study will be carried out at Multidisciplinary Pain Centre, Rigshospitalet, investigating opioid treated chronic non-cancer patients. These patients should have been treated only with one opioid for more than one month and will be compared to an age, educational and sex matched control group of chronic non-cancer patients not treated with analgesics.

STUDY SAMPLE

The study is an explorative study of 25 opioid treated patients and 25 controls.

The patients will be included or excluded for either group on the basis of specific criterions.

If the hypotheses of the study seem to be confirmed more patients will be included in order to investigate the effects of different opioid substances.

METHOD

Data will be collected by a trained medical student, who will administer the instruments and retrieve information from the patients' files.

Hormone assay

The adrenocortical function will be tested with the 30 min ACTH test. Leydig-cell function, IGF, TSH, thyroxine and prolactine will be measured as well.

Immunology Fresh whole blood will be used for flow cytometry, where the amount of the different cells in the immune system will be measured. Furthermore, plasma samples (snap frozen) will be collected (biobank).

The following cell types will be analyzed by using flow cytometry: NK cells, B cells and T cells. To study the immune response fresh whole blood will be stimulated with pathogens. Production of cytokines will be examined by analyzes of culture supernatants. Possible alteration in inflammation will be determined by analysing the plasma samples.

Establishment of research biobank

All material is collected as part of the study. A biobank will be established and blood samples will be safely stored at Rigshospitalet as long as the study is going on. The purpose of the research biobank is to use the samples in follow-up studies.

Assessment of cognitive function

Regarding neuropsychological assessment, two instruments were selected:

1. CRT measures sustained attention or vigilance. It is a computer test, in which through headphones, 100 auditory signals are delivered to the patient at random intervals. The patient is instructed to press a button as soon as the sound is heard.
2. DST assesses attention/concentration, recent and working memory. Patients are asked to repeat the series of numbers of increasing lengths, in both forward (direct) and backward (reverse) order.

Pain evaluation

Patients' pain intensity will be assessed using the Brief Pain Inventory (BPI) measuring pain at its worst, least and average during the last 24 hours and the current pain intensity.

Mood

Depression and anxiety will be evaluated using the Hospitality Anxiety and Depression Scale (HADS). Scores above 8 indicates that a depressive or anxiety disorder is likely to be present.

Health-related quality of life

The Short Form 36 (SF-36) will also be included in the self-administered questionnaire. The SF-36 is a 36-item survey that measures eight dimensions of health. Higher scores on the SF-36 (range 0 to 100) indicate better health-related quality of life.

RESULTS

The results will be analysed by using specific statistic tools as descriptive variables, primary outcome, secondary outcome, significance levels, and clinical significance.

ELIGIBILITY:
CRITERIA FOR INCLUSION IN THE OPIOID GROUP

* Age >18 yrs and <65 yrs
* Chronic non-cancer pain (>6 months' duration)
* At least six years of schooling
* Fluent in spoken and written Danish
* On opioid treatment (>30 mg of morphine equivalents pr. day) for at least one month

CRITERIA FOR INCLUSION IN THE CONTROL GROUP

* Age >18 yrs and <65 yrs
* Chronic non-cancer pain (>6 months' duration)
* At least six years of schooling
* Fluent in spoken and written Danish (no need for translator)
* No analgesic treatment for the last month

CRITERIA FOR EXCLUSION

* Treatment with glucocorticoid or sex hormones within the previous 6 months or on-going therapy with drugs known to interfere with endocrine function
* Treatment with adjuvant analgesics (anticonvulsants, antidepressants and others), NSAIDs/paracetamol, benzodiazepines and hypnotics (sleeping pills can be discontinued 3 days before testing) the last month
* Known endocrine disease including insulin treated diabetes mellitus
* Previously diagnosed dementia or encephalopathy
* Brain trauma necessitating hospitalization within last 6 months
* Previously diagnosed liver disease
* Renal insufficiency (serum creatinine concentration >140 µmol/l)
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pain patients at Multidisciplinary Pain Centre at Rigshospitalet, Denmark
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
Dose and time dependent effects | Up to 2.5 years
  Differences on the mean results of endocrine and immunologic blood tests between patients and controls, considering dose and time dependent effects.

SECONDARY OUTCOMES:
Function of the immune and endocrine systems | Up to 2.5 years
  Differences on the mean scores of the cognitive tests, pain intensity and quality of life between patients and controls.

CONTACTS AND LOCATIONS:
Overall Officials: Per Sjøgren, Proff., Principal Investigator — Rigshospitalet, Denmark